# Statistical Analysis Plan

Observational study Protocol

EMR 700623-545

Identification No.

Title: A Phase IV, prospective, randomized, exploratory,

multicenter, Eeva trial (Time Lapse Eeva - TiLE)

**Observational study Protocol** 

Version 4.0/12 February 2015

Version/Date

Statistical Analysis Plan Author

PD PD

Statistical Analysis Plan

20FEB2017/ Version 1.0

**Date and Version** 

**Statistical Analysis Plan Reviewers** 



- , Study Statistician
- 2. PPD , Biostatistician
- 3. PPD , Principal Biostatistician

# **Merck Serono**

- 1. PPD , PPD
- 2. PPD
- 3. PPD

### Confidential

This document is the property of Merck KGaA, Darmstadt, Germany, or one of its affiliated companies.

It is intended for restricted use only and may not - in full or part - be passed on, reproduced, published or used without express permission of Merck KGaA, Darmstadt, Germany or its affiliate.

Copyright © 2017 by Merck KGaA, Darmstadt, Germany or its affiliate. All rights reserved.

# 1 Signature Page

Statistical Analysis Plan: EMR 200623-545

A Phase IV, prospective, randomized, exploratory, multicenter, Eeva trial (Time Lapse Eeva – TiLE)



# 2 Table of Contents

| 1 | Signature Page | 2 |
|--------|---------------------------------------------------------------|----|
| 2 | Table of Contents | 3 |
| 3 | List of Abbreviations and Definition of Terms | 5 |
| 4 | Purpose of the Statistical Analysis Plan | 6 |
| 5 | Summary of Clinical Study Features | |
| 5.1 | Primary endpoint | 6 |
| 5.2 | Secondary endpoints | 6 |
| 5.3 | Selection of Trial Population and randomization | 6 |
| 5.4 | Documented variables | |
| 5.4.1 | Screening and treatment | 6 |
| 5.4.2 | Oocyte Retrieval | |
| 5.4.3 | Embryo Day 3 | 7 |
| 5.4.4 | Embryo Transfer | |
| 5.4.5 | Embryo Day 5-6 | 7 |
| 5.4.6 | Dates | |
| 5.4.7 | Post Oocyte Retrieval or Post Transfer Day 12-18 | 7 |
| 5.4.8 | Gestational Age Week 5-8 (Transfer and Treatment Outcome | |
| | eCRF) | 7 |
| 5.4.9 | Post-Pregnancy follow-up | |
| 5.4.10 | Additional Ultrasound > 8 weeks (Optional) | |
| 5.4.11 | Assessment of Safety | |
| 6 | Sample Size/Randomization | 8 |
| 7 | Overview of Planned Analyses | |
| 7.1 | Sequence of Analysis | |
| 7.2 | Interim Analysis. | 8 |
| 7.3 | Final Analysis | 8 |
| 8 | Analysis Sets | 8 |
| 8.1 | Intention-to-treat (Full Analysis Set) | 8 |
| 8.2 | Subgroups EC and ENC within the Eeva plus morphology | |
| | grading group | 8 |
| 8.3 | Added selection | |
| 9 | General Specifications for Statistical Analyses | 9 |
| 10 | Study Subjects | |
| 10.1 | Disposition of Subjects and Discontinuations | |
| 10.2 | Protocol Deviations | 9 |
| 11 | Demographics and Other Baseline Characteristics | 9 |
| 11.1 | Demographics, Medical History, Other Baseline Characteristics | 9 |
| 11.2 | Descriptive tables for post-baseline variables | |
| 12 | Previous or Concomitant Medications/Procedures | |
| 13 | Treatment Compliance and Exposure | 10 |
| 14 | Endpoint Evaluation | |

| 14.1 | Primary analysis | 10 |
|---------|--------------------------------------------|----|
| 14.2 | Implantation rate in other selections | 10 |
| 14.3 | KID selection | 10 |
| 14.4 | Secondary variables selection of ITT | 10 |
| 14.5 | Secondary variables KID | 10 |
| 14.6 | Exploratory Variables | |
| 15 | Safety Evaluation | 12 |
| 16 | References | 12 |
| 17 | Used Variables | 12 |
| 18 | Table description: principles of reporting | 15 |
| 18.1 | Generalities | |
| 18.1.1 | Type of table | 15 |
| 18.1.2 | Format | |
| 19 | List of Tables of the report | 15 |
| 19.1 | Randomization | |
| 19.2 | Screening | 16 |
| 19.2.1 | Inclusion/exclusion: | 16 |
| 19.2.2 | Patient Disposition | 16 |
| 19.2.3 | Comparison at baseline | 16 |
| 19.2.4 | Treatment | 16 |
| 19.2.5 | Oocytes Retrieval | 16 |
| 19.2.6 | Transfer | 16 |
| 19.2.7 | Additional Optional Ultrasound | 17 |
| 19.2.8 | device Incident | |
| 19.2.9 | Study Exit | 17 |
| 19.2.10 | Dates | 17 |
| 19.2.11 | Safety | |
| 20 | Table format | 18 |

# 3 List of Abbreviations and Definition of Terms

AE Adverse Event

BP Biochemical Pregnancy

CP Clinical Pregnancy

CPR Clinical Pregnancy Rate

EC Eeva Conform

Eeva Early embryo Viability Assessment

EMG arm treated Eeva + Morphology grading

ENC Eeva Non-conform

IR Implantation Rate

ITT Intent to Treat

KID Known Implantation Data

MG arm Morphology Grading only

MP Multiple Pregnancy

nET Number of Transferred Embryos

nFS Number of Foetal Sacs

OP On Going Pregnancy

**OPR** Ongoing Pregnancy Rate

RR Risk Ratio

SM Spontaneous Miscarriage

SMR Spontaneous Miscarriage Rate

TRT Treatment Variable

**UR** Utilization Rate

# 4 Purpose of the Statistical Analysis Plan

Eeva is a time lapse monitoring system able to picturing embryos every 5 minutes during embryo culture and embryo development. The standard technique (Morphology Grading MG) is based on multiple observations of embryos under regular light microscopes, known of limited predictive value: In a Trial, from 2 embryos chosen by MS, 39%, 38% and 23% of cycles resulted in none, one and two blastocysts, respectively. The benefits demonstrated during the first investigations of Eeva is a specificity of 85%. (Eeva should detect 85% of transferred failed embryos). The purpose of this plan is the evaluation of the Early Embryo Viability Assessment (Eeva) efficacy in predicting confidence intervals for relative embryo implantation potential over baseline outcomes

# 5 Summary of Clinical Study Features

### 5.1 Primary endpoint

The primary objective of the trial is the point and relative interval estimate of the Implantation Rate (IR) performed on day 3 or day 5 (with and without genetic analysis) in the groups Eeva plus MG (EMG) and MG alone (MG)

## 5.2 Secondary endpoints

- (a) Utilization Rate (UR) (number of transferred and frozen embryos divided by number of normally fertilized oocytes x 100),
- (b) Clinical Pregnancy Rate (CP) (assessed by ultrasonography at weeks 5 to 8),
- (c) Ongoing Pregnancy Rate (OP) (assessed by ultrasonography at weeks 10 to 12),
- (d) Multiple Pregnancy Rate (MP) (assessed by ultrasonography at weeks 5 to 8) and
- (e) Spontaneous Miscarriage (SM).
- (e) Drugs protocol type (GnRH agonist/GnRH antagonist) and gonadotrophin dose for Controlled Ovarian Stimulation in relation with Eeva categories and implantation outcomes.
- 5.3 Selection of Trial Population and randomization

See protocol section 5.3 and 5.6

#### 5.4 Documented variables

#### 5.4.1 Screening and treatment

Inclusion Criteria, Age, Pregnancy History, Number of attempts, Number of Spontaneous abortions, Number of Live Births, Number of Non-ART cycles, Number of Fresh ART cycles, Number of Frozen ART cycles, Follicle Stimulating Hormone Maximum, Follicle Stimulating Hormone Units, Anti Mullerian Hormone Max, Anti Mullerian Hormone Unit, Estradiol Max, Estradiol Units, Luteinizing Hormone Max, Luteinizing Hormone Units, Antral Follicle Count,



Male Infertility, Polycistic Ovaries, Reduced Ovarian Reserve, Tubal Factor, Unexplained, Other.

Treatment variables: Protocol of Stimulation, stimulation medication, Time of hCG trigger to oocyte retrieval, Pre-trigger Endometrium (Trt Set).

### 5.4.2 Oocyte Retrieval

Number of oocytes retrieved; Andrology information; Insemination method; Total number of normally fertilized eggs (2PN); Culture conditions (including gas phase, media, and protein, etc.); Embryo morphological grading may be assessed on Day 2 as per local laboratory standard practice in those subjects randomized to the Morphology group only.

#### 5.4.3 Embryo Day 3

Type of Eeva Petri Dish (number of micro-wells); Eeva micro-well identification; Cell stage and Morphology grading; Eeva results; Fate of each embryo (Transferred, Cryopreserved, Discarded or extended culture to Day 5/6); Eeva Petri Dish and Scope information; Culture conditions.

#### 5.4.4 Embryo Transfer

Date and day of transfer; Luteal phase support; Use of ultrasound; Final number of embryos transferred.

#### 5.4.5 Embryo Day 5-6

Type of Eeva Petri Dish (number of micro-wells); Eeva micro-well identification; Development stage and Morphology grading; Fate of the embryo (Transferred, Cryopreserved, Discarded or extended culture to Day 5/6); Eeva Petri Dish and Scope information; Culture conditions

### 5.4.6 Dates

All date of each stage are available

# 5.4.7 Post Oocyte Retrieval or Post Transfer Day 12-18

Pregnancy test results, Quantitative hCG, as applicable. If the result of the pregnancy test is negative, the subject will have completed the trial and be exited at that time.

# 5.4.8 Gestational Age Week 5-8 (Transfer and Treatment Outcome eCRF)

Result of initial pregnancy ultrasound; Number of intrauterine gestational sacs; Number of fetal heartbeats. If the result of the ultrasound is negative (no fetal heartbeat is detected), the subject stops



# 5.4.9 Post-Pregnancy follow-up

Pregnancy outcome

### 5.4.10 Additional Ultrasound > 8 weeks (Optional)

Result of initial pregnancy ultrasound; Number of fetal sacs and number of fetal heartbeats

# 5.4.11 Assessment of Safety

Safety of Eeva will be evaluated by assessment of device deficiency only. Each individual occurrence will be listed.

# 6 Sample Size/Randomization

See protocol 5.3

# 7 Overview of Planned Analyses

## 7.1 Sequence of Analysis

One sequence

#### 7.2 Interim Analysis

Interim analysis was planned when half of the patients completed the study in the protocol. But based on medical affairs advice it was decided not to conduct the interim analysis.

### 7.3 Final Analysis

See section 8 below

### **Changes to the Planned Analyses**

No changes

### 8 Analysis Sets

The following sets of subjects will be considered in the analysis:

#### 8.1 Intention-to-treat (Full Analysis Set)

The intention-to-treat population includes all randomized subjects. Due to the fact that this is an exploratory trial in contrast to usual definitions of ITT ('presented as randomized') subjects will be presented based on the method used (EvMG = Eeva scores plus morphology grading, MG=morphology grading only).

# 8.2 Subgroups EC and ENC within the Eeva plus morphology grading group

The EEVA Time Lapse system assists the embryologist in improving embryo assessment accuracy. Whether the embryologist follows the recommendation made by the system is the decision of the embryologist. Therefore two subgroups will be considered:



- (a) Subjects form Eeva scores plus morphology grading group for whom the embryologist has followed the recommendation of the Eeva system (group noted EC or Eeva conform). As the principle selection algorithm for the test arm of the study the selection of embryos for transfer is based on the recommendations made by the EEVA system.
- (b) Subjects form Eeva scores plus morphology grading group for whom the embryologist has NOT followed the recommendation of the Eeva system (group noted ENC or Eeva Not conform). Every effort at the site will be made to keep this case to a minimum of cases as investigators are encouraged to use their technical expertise and follow the EEVA system recommendations. However, on investigators' discretion and patients' best interests it may be decided to exceptionally disregard the system recommendation when such recommendation contradicts the morphological pre-assessment of the embryos.

will share the "Embryo Days 2, 3, 5, 6 Laboratory Data Morphological/EEVA Grading" data with Merck after the database lock.

#### 8.3 Added selection

The KID sample (Known Implantation Data) is the subset of ITT sample such that the IR=0% or 100% (for single,double or triple) mbryo transfer, ITT=KID; for other implantations, women such that 0<IR<1<2<3 will be disregarded).

### 9 General Specifications for Statistical Analyses

# 10 Study Subjects

### 10.1 Disposition of Subjects and Discontinuations

This table will provide the distribution of the randomized patients for each group into completers and non completers. For completers, the table will provide the distribution of the type of completion (variable cycleCST, cfr section 19), and for non completers, the distribution of the reason of non completion (variable cycleNST, cfr section 19).

# 10.2 Protocol Deviations

Protocol deviations will be determined before database lock.

## 11 Demographics and Other Baseline Characteristics

# 11.1 Demographics, Medical History, Other Baseline Characteristics

Table will describe each group EMG and MG on all the above described existing variables at baseline. Depending on the type of variable, two-way Crosstab or Mean tables across (EMG/MG) Groups will be provided (cfr table contents and individual description of these tables in section 19).

#### 11.2 Descriptive tables for post-baseline variables

For all the variables after baseline, each variable (described in table 19) will be documented for each subgroup (EMG/MG) according a frequency two-way cross tabulation or a mean table, depending on the type of variable (nominal, continuous).



# 12 Previous or Concomitant Medications/Procedures

Does not apply

### 13 Treatment Compliance and Exposure

Does not apply

## 14 Endpoint Evaluation

### 14.1 Primary analysis

Implantation rate will be analyzed with two definitions

First definition: The IR (at embryo level) corresponding to a group of patients is calculated as the ratio of the total fetal sacs (nFS) identified by ultrasonography at weeks 5 to 8 divided by the number of embryos transferred (nET), thus IR=nFS/nET.

Alternative Definition of Implantation Rate: The previous (and usual) calculation of IR as mentioned in the protocol (IR=nFS/nET) has problems, in particular the implanted embryos are not independent. The international definition used by WHO in particular (see for instance <a href="http://www.advancedfertility.com/ivf.htm">http://www.advancedfertility.com/ivf.htm</a>) is: The alternative definition IR\* at women level is  $IR_w = nFS_w/nET_w$  and  $IR^* = (1/n)$ .  $\Sigma_{w=1,n} IR_w$ .

Note: The two definitions IR and IR\* coincide in some cases, in particular for elective Single Embryo transfer eSET (where only one embryo is transferred) or when KID sample is used, but in the general case (ITT sample for instance, IR and IR\* will be different).

The point estimate and 95% CI of IR and IR\* will be calculated in both groups EMG and MG for the ITT selection. No inferential comparison will be conducted between these two groups (as this study is purely descriptive).

The following sections are considered as secondary analyses.

### 14.2 Implantation rate in other selections

The point estimate and 95% CI of IR and IR\* will be calculated in the subgroups EC and ENC. No tests of comparison between any subgroup will be conducted.

### 14.3 KID selection

The same calculations will be conducted for EMG and MG groups and EC and ENC restrained to KID selection.

### 14.4 Secondary variables selection of ITT

Utilization Rate (UR), Clinical Pregnancy rate (CP), Ongoing Pregnancy rate (OP), Multiple Pregnancy rate (MP), Spontaneous Miscarriage (SM). The estimate and 95% CI will be calculated in both groups EMG and MG, and in both groups EC and ENC.

#### 14.5 Secondary variables KID

The same analysis will be conducted on KID selection for Utilization Rate (UR), Clinical Pregnancy rate (CP), Ongoing Pregnancy rate (OP), Multiple Pregnancy rate



(MP), Spontaneous Miscarriage (SM) . The estimate and 95% CI will be calculated in both groups EMG and MG, and in both groups EC and ENC.

# 14.6 Exploratory Variables

Multiple Linear regression analysis of IR (based on subject level) as dependent variable and treatment as independent parameter effected by the following confounding factors

| Factors | Description |
|---|---|
| Stimulation protocol | Categorical variable, 3 states: Agonist Luteal phase;<br>Antagonist; and Agonist Mirco-dose Flare and Other |
| Drugs used | Categorical variable, 3 states: recombinant Gn, urinary Gn, and mix-use of recombinant and urinary Gns |
| Day of transfer | Categorical variable, 2 states: D3 Vs D5/6 |
| Age of patients | Continuous variable, years |
| Culture<br>medium | Categorical variable, 5 states: Quinn's Advanced Fertilization,<br>Global Medium, Vitro life G-IVF, Irvine Single Step<br>Medium, and Other |

A better estimate of implantation rate will be obtained based on subject level adjusted for confounding factors by a Multiple Linear regression.

Given the exploratory nature of the design, the model will be investigated stepwise and repeated backward. The final model will exclude backward P-values > 0.10.

The Center effect will also to be considered in the model.

The results of regression analysis will be reported with the following items

- ➤ Regression Coefficient with 95% CI
- Standard Error
- > P-value
- ➤ Coefficient of Determination (R<sup>2</sup>)

# **Subgroup analyses**

Further subgroup analysis based on selected baseline parameter could be conducted as follows.

1) IR of the two treatment groups at each site (descriptive summary statistics with 95% CI,



and RR with 95% CI and P value). The Risk Ratio, 95% CI and P-value will be calculated, provided the number of subjects in a site will be at least 30, otherwise only descriptive statistics will be provided for that particular site.

- 2) IR, CPR, OPR and SMR of the two treatment groups for subgroups of patients with ET on D3 and D5/6 (descriptive summary statistics, RR with 95% CI and *P* value);
- 3) IR, CPR, OPR and SMR of the two treatment groups for subgroups of patients with age ≤35 and >35(descriptive summary statistics, RR with 95% CI and P value).
- 4) IR of the two treatment groups for subgroups of patients using 5 types of culture media (descriptive summary statistics, RR with 95% CI and *P* value).
- 5) IR of subgroups of patients using 5 types of culture media (regardless the method of embryo assessment, descriptive summary statistics and 95% CI)

# 15 Safety Evaluation

In conformity with protocol, device deficiency will be individually listed.

#### 16 References

No reference at this stage

#### 17 Used Variables

In the following table, each variable is characterized by its ID (short name), variable label, type (B=Binary, I=Numerical Integer (such as count), C=Categorical, F=Real Numeric). Format (I.J where I denotes the total number of digits, and J=number of decimals, i:j is a format with j decimals for the tables, but 0 decimal for data list, while i.j denotes j decimals for the tables and data list). The groups of binary variables highlighted in gray will be presented on the same table.

| <u>Variable</u><br><u>ID</u> | Variable Label | Type | <u>Fmt</u> | Value Labels |
|---|---|---|---|---|
| Baseline Va | ariables | | | |
| Inc<1,13> | Inclusion Criteria | В | | |
| Age | Age | I | 6:1 | |
| Preg1 | Pregnancy History | В | | |
| Preg2 | Number of attempts | ı | 6:1 | |
| Preg3 | Number of Spontaneous abortions | I | 6:1 | |



| Preg4 | Number of Live Births | I | 6:1 | |
|---|---|---|---|---|
| Pt1 | N of Non-ART cycles | ı | 6:1 | |
| Pt2 | N of Fresh ART cycles | I | 6:1 | |
| Pt32 | N of Frozen ART cycles | I | 6:1 | |
| FSHm | Folicle Stim Hormone<br>Maximum | F | 8.2 | |
| FSHu | Folicle Stimulating Hormone Units | F | 8:2 | |
| AMHm | Anti Mullerian Hormone Max | F | 8.2 | |
| AMHu | Anti Mullerian Hormone Unit | F | 8:2 | |
| E2m | Estradiol Max | F | 8.2 | |
| E2u | Estradiol Units | F | 8:2 | |
| LHm | Luteinizing Hormone Max | F | 8.2 | |
| LHu | Luteinizing Hormone Units | F | 8:2 | |
| AFC | Antral Follicle count | I | 6:1 | |
| RI1 | Male Infertility | В | | |
| RI2 | Polycistic Ovaries | В | | |
| RI3 | Reduced Ovarian Reserve | В | | |
| RI4 | Tubal Factor | В | | |
| RI5 | Unexplained | В | | |
| RI6 | Other | В | | |
| Prot | Stimulation protocol | С | 4 | 1=Agonist Luteal Phase Start 2=Agonist Micro-Dose Flare 3=<br>Antagonists suppression 4=Other |
| FSHtd | rFSH (Total Dose) | F | 8.2 | |
| FSHnd | rFSH (N of Days) | F | 8:2 | |
| LHtd | rLH (Total Dose) | F | 8.2 | |
| LHnd | rLH (N of Days) | F | 8:2 | |
| FLtd | rFSH-rLH (Total Dose) | F | 8.2 | |
| FLnd | rFSH-rLH (N of Days) | F | 8:2 | |
| Hmgtd | Hmg (Total Dose) | F | 8.2 | |
| Hmgnd | Hmg (N of Days) | F | 8:2 | |
| Ufshtd | uFSH (Total Dose) | F | 8.2 | |
| Ufshnd | uFSH (N of Days) | F | 8:2 | |
| Ottrttd | Other treatments (Total Dose) | F | 8.2 | |
| ottrtnd | Other treatments (N of Days) | F | 8:2 | |
| stimdur | Total number of days of stimulation | I | 8:2 | |

| E2pk | Peak estradiol | F | 8.2 | |
|---|---|---|---|---|
| E2u | Unit Estradiol | В | 4 | 1=pmol/L 2=pg/mL |
| Nfol12 | N of follicles > 12mm | I | 5:1 | |
| Nfol18 | N of follicles > 18 mm | I | 5:1 | |
| endoth | Endometrium Thickness | F | 8.2 | |
| Post Basel | <br> ine Variables | | | |
| Noo | N of oocytes | I | 8:1 | |
| Noom | N of Mature oocytes | I | 8:1 | |
| Sps | Sperm Sample | С | 4 | 1=Fresh 2=Frozen 3=both |
| Itype | Insemination Type | С | 4 | 1=ICSI 2=Ivf 3= Both |
| Cult | Culture medium | С | 4 | 1= Quinns Advantage Fertilization 2= Global Medium 3= Vitrolife<br>G-IVF 4= Irvine Single Step Medium 5= Other |
| Incub1 | Incubator Information O2 | С | 4 | 1= 5% 2=20% |
| Incub2 | Incubator CO2 | F | 8.2 | |
| Psupp | Protein Supplement | С | 4 | 1= None used, 2 = SPS, 3 = HAS, 4 = SSS, 5 = Other |
| Negg | N of retrieved eggs | I | 6.1 | |
| eggGV | Egg type GV | В | | |
| eggMI | Egg type MI | В | | |
| eggMII | Egg type MII | В | | |
| eggOt | Egg type Other | В | | |
| Trf | Was a transfer attempted ? | В | | |
| Nte | N of transferred Embryos | I | 4.1 | |
| Usg | Ultra sound guided | В | | 1=Yes 2=No |
| Cat1 | Catheter Typ Mucous | В | | |
| Cat2 | Catheter Typ Blood | В | | |
| Cat3 | Catheter Typ retained embryos | В | | |
| Cat4 | Catheter Typ N/A | В | | |
| Grading | Procedure Grading | С | 4 | 1= Easy 2= Difficult |
| Pdg | Embryo assessed by PGD/PGS | С | 4 | 1=Yes 2=No |
| Euploid | Euploid transferred ? | В | 4 | |
| LPS | Luteal Phase support | В | | 1=Yes 2=No |
| DelMet | Delivery Method | С | | 1= Crinone 2=Endometrin 3=Other Vaginal 4=Intramuscular 5=Other |
| Test1 | Post Transfer test 1 | В | | 1= Urine 2=Blood |
| Test1r | Post Transfer test 1 result | В | | 1= Positive 2= Negative |
| Test2 | Post Transfer test 2 | В | | 1= Urine 2=Blood |
| Test2r | Post Transfer test 2 result | В | | 1= Positive 2= Negative |

| US1 | Ultra Sound result | В | | 1= Positive 2= Negative |
|---|---|---|---|---|
| Nsac | N of gestational Sacs | ı | 4:1 | |
| Nhbt | N of Heartbeats | I | 4:1 | |
| Outc | Final outcome further to Ultra<br>Sound | С | | 1=No pregnancy 2=Biochemical pregnancy 3=Ectopic<br>4=miscarriage 5= Ongoing |
| EndPP | Cycle completed on Per<br>Protocol | В | | 1=yes 2=o |
| cycleCSt | IF cycle complete : Status | С | | 1= Ongoing pregnancy 2= Pregnancy came to term 3= Pregnancy lost 4= Failed to conceive 9= therapeutic abortion 10= Other |
| cycleNst | If cycle non complete : Status | С | | 0=Normal 1= OHSS risk 2= Embryo transfer cancelled 5= Freeze all<br>6= Other 7= Imaging discontinued prior to completion 8= Subject<br>requested to be withdrawn 9= Investigator withdrew subject 10=<br>Subject was lost to follow-up 11= Subject was noncompliant |

# 18 Table description: principles of reporting

### 18.1 Generalities

Unless otherwise specified, all these tables are two-way table in subdividing the whole sample following treatment group (trt).

# 18.1.1 Type of table

DataList Individual list of a subset of variables in text format for a selection of patients Mean Mean, SD, Count, Minimum, Maximum, quartiles (ex: Section 20, table 1)

Mean, SD, 95%CI, count (ex: Section 20, table 2)

Perc Percentage, Count (ex : Section 20, table 3)

PercCl Percentage, Count, 95% Cl (ex : Section 20, table 4)

CrossTab Two-way Cross-tabulation with count and % in columns (ex : Section 20, table 5)

# 18.1.2 Format

| Percentage and associated CI | 1 decimal |
|---|---|
| Proportion | 3 decimals |
| Count | 0 decimals |
| Continuous variable described by mean, quartiles, range, standard deviation and their CI | Conform to goldilocks rounding ref: Lang T, Altman D. Basic statistical reporting for articles published in clinical medical journals: the SAMPL Guidelines. (cited 19 June 2014). http://www.equator-network.org/wp-content/uploads/2013/07/SAMPL-Guidelines-6-27-13.pdf |

# 19 List of Tables of the report

## 19.1 Randomization



Data List with Patient ID, randomization Date, Treatment code 0=MG, 1=EMG

## 19.2 Screening

### 19.2.1 Inclusion/exclusion:

Data List ID patients list out of exclusion/inclusion criteria

Cross-tab Inclusion/exclusion by TrT

### 19.2.2 Patient Disposition

crossT cycleST \* trt
crossT cycleNST \* trt

### 19.2.3 Comparison at baseline

Mean Age \* trt

Mean Number of pregnancies, Abortions, Live Births \* trt
Mean Number of Gonad cycles, Fresh , Frozen Art Cycles \* trt

Mean FSH, AMH, E2, LH, AFC (units/ Maximum) \* trt

CrossT Reason for ART \* trt

### 19.2.4 Treatment

CrossT Stimulation Protocol \* trt

Mean rFSH, rLH, rFSH+rlH,hMG, uFSH \* trt
Mean Thickness of endometrium \* trt

### 19.2.5 Oocytes Retrieval

Mean NOO, NMO \* trt

Mean Sperm \* trt

CrossT Type of Insemination \* trt
CrossT culture Medium \* trt

Mean CO2, O2 \* trt (Incubator information)

Mean Total Number of Eggs \* trt

### 19.2.6 Transfer

Percent Transfer (0/1) \* trt

Percent conformity with Eeva \* trt

Percent nET \* trt

Percent Ultrasound guided \* trt
DataList Brand of Ultrasound
crossT Catheter Type \* trt

CrossT Grading of Procedure \* trt

Percent embryos assessed with PDG

Percent euploid Transformed
Percent Luteal Phase provided
crossT method of delivery
crossT Urine Sample-A/B \* trt
crossT Urine-A/B-Result \* trt
mean Quant-HCG-A/B \* trt

Percent (InitialPregnancyUS, nFS, nHeartBits) \* trt

# 19.2.7 Additional Optional Ultrasound

Percent (InitialPregnancyUS, nFS, nHeartBits) \* trt (for

# 19.2.8 device Incident

DataList Patient, Time, Eeva component, Description, troubleshooting, contact

# 19.2.9 Study Exit

CrossT Study exit Categories \* trt

# 19.2.10 Dates

data list for each patient, the dates associated with each event (from Recruitment to Live birth)

# 19.2.11 Safety

Each Individual device deficiency event will be listed.

# 20 Table format

| | Mean | SD | Q1 | Median | Q3 | Min | Max | Count |
|---------|------|------|------|--------|------|------|-------|-------|
| MG | 3.68 | 2.82 | 2.00 | 3.00 | 5.00 | 0.00 | 13.00 | 155 |
| Eeva+MG | 3.28 | 2.59 | 1.00 | 3.00 | 5.00 | 0.00 | 11.00 | 142 |
| Total | 3.49 | 2.72 | 1.00 | 3.00 | 5.00 | 0.00 | 13.00 | 297 |

Table 1. example of a Mean table

| | Mean | 95% CI | Count |
|---------|------|------------|-------|
| MG | 3.57 | 3.12, 4.01 | 143 |
| Eeva+MG | 3.40 | 2.91, 3.88 | 124 |
| Total | 3.49 | 3.16, 3.81 | 267 |

Table 2. example of a Mean table with 95%CI

| | Percent | Count |
|---------|---------|-------|
| MG | 12.6 | 135 |
| Eeva+MG | 9.6 | 135 |
| Total | 11.1 | 270 |

Table 3. example of a Percent table

| | Percent | 95% CI | Count |
|---------|---------|-------------|-------|
| MG | 13.9 | 8.56, 20.81 | 137 |
| Eeva+MG | 6.7 | 3.11, 12.37 | 134 |
| Total | 10.3 | 6.97.14.59 | 271 |

Table 4. example of a Percent table with 95%CI

| | MG | | Eeva+MG | | Total | |
|-------|-------|-------|---------|-------|-------|-------|
| | Count | Col % | Count | Col % | Count | Col % |
| GBR | 4 | 2.9 | 8 | 5.9 | 12 | 4.4 |
| HUN | 7 | 5.1 | 12 | 8.9 | 19 | 7.0 |
| LVA | 7 | 5.1 | 12 | 8.9 | 19 | 7.0 |
| SWE | 1 | 0.7 | 0 | 0.0 | 1 | 0.4 |
| Total | 137 | 50.4 | 135 | 49.6 | 272 | 100.0 |

Table 5. example of a Cross table (Count, Col %).